## Project Protocol

# Improvement of Patient Satisfaction and Clinical Outcomes Using JointCOACH to Manage the Episode of Care for THA and TKA Bundles

Principle Investigator: Carlos Higuera, MD

Research Program Manager: Alison Klika, MS

Research Coordinator: Anabelle Visperas, PhD

## **Table of Contents:**

| 1. | Project Summary | 3 |
|----|------------------------------------------|------|
| 2. | Introduction and Background | 3 |
| 3. | Specific Aims | 4 |
| 4. | Methods | 5 |
| | 4.1 Study Design | 5 |
| | 4.2 Patient Population | 6 |
| | 4.3 Sample Size Calculation | 7 |
| | 4.4 Schedule of Events. | 8 |
| | 4.5 Data Analysis | 9 |
| 5. | References | . 10 |
| 6. | Appendix | 11 |
| | 6.1 Study Metrics | . 11 |
| | 6.2 ICD-10 codes for relevant metrics | . 12 |
| | 6.3 Success Thresholds for Study Metrics | . 13 |
| | 6.4 Provider Satisfaction Survey | . 14 |

#### 1. Project Summary

JointCOACH is a web-based communication platform that enables joint replacement patients to communicate with their care team via computer or smartphone throughout their episode of care, from the time that surgery is scheduled until at least 90 days postoperatively. Patients will receive the following information at key intervals: 1) instructions about how to prepare for surgery, 2) information about the procedure, 3) information about medications and pain control, 4) information about postoperative recovery and rehabilitation. In addition, several surveys will be distributed using JointCOACH to keep patients involved in their own recovery and to keep the surgical team informed of their progress. The proposed research will help determine if JointCOACH can improve patient satisfaction and clinical outcomes.

## 2. Introduction and Background

Health systems invest significant resources to improve quality and reduce costs. However, this process is typically driven by hospital administration and staff. Recently, studies have shown that when patients are engaged, they take more responsibility for their own health and preventative care. Additionally, these patients are more satisfied with their healthcare experiences and have lower rates of healthcare utilization <sup>1,2</sup>. Physicians are in the best position to promote patient engagement since they have direct relationships with their own patients. However, physicians need frictionless tools with minimal implementation barriers in order to create and maintain this relationship in the follow up period.

Patient engagement has been referred to as the next blockbuster "drug", and increasing evidence demonstrates that highly engaged patients not only enjoy improved outcomes, but have fewer complications, undergo fewer readmissions, and have lower total costs of care <sup>3–5</sup>. While these engagement-related outcomes have been shown in several other specialties, relatively little has been done to explore this relationship in orthopedics. The opportunity to demonstrate the

impact of engagement on outcomes in the orthopedic space is highlighted by the estimated \$1.5B of medical expenses occurring nationally due to potentially preventable readmissions following orthopedic surgeries alone.

Stryker Performance Solutions JointCOACH<sup>TM</sup> and the Cleveland Clinic are interested in collaborating on a clinical pilot study to demonstrate that high patient engagement leads to enhanced preoperative preparation potentially reducing length of stay (LOS), readmissions and reoperations, increasing discharge disposition to home rather than another facility, reducing the need for in-person follow up, and increasing patient (and provider) satisfaction after elective primary hip and knee arthroplasty (THA and TKA). These improvements can translate to higher financial savings through the episode of care especially in light of the alternative payment models.

## 3. Specific Aims

Currently in use by orthopedic groups around the country, JointCOACH improves perioperative outcomes after THA and TKA and mitigates risk by: 1) enhancing patient engagement with providers, 2) allowing patients to play an integral role in patient-reported outcomes, 3) generating and relaying actionable pre- and postoperative reporting directly to the clinical team, and 4) detecting impending postoperative complications early, enabling timely intervention and preventing avoidable complications and readmissions. The specific aims of this proposal are to:

- 1. Measure patient satisfaction with and without use of JointCOACH as a tool for patient engagement
- 2. Understand the degree to which high postoperative engagement can reduce the amount of healthcare resource utilization by answering the following questions:

- a. Will the use of JointCOACH decrease the number of potentially avoidable healthcare utilization encounters such as Emergency Department (ED) and hospital visits (i.e. readmissions and reoperations)?
- b. Does utilizing JointCOACH improve clinical workflow by minimizing telephone calls and thereby offloading support staff, allowing them to be more efficient?
- c. Does utilizing JointCOACH reduce the volume of on-call pages by addressing patient questions up front, alleviating concerns, and providing them with the information they need when they need it?
- d. Does utilizing JointCOACH allow the practice to identify patients whose in-person follow-up needs are minimal?
- 3. Measure additional potential benefits including shorter length of hospital stay, discharge disposition to home rather than a facility and decreased 90 day readmissions and reoperations by answering the following:
  - a. Does utilizing JointCOACH lead to early detection of adverse signs/symptoms that develop between clinical encounters and result in reduced readmissions and reoperations?
- 4. Evaluate the financial impact of JointCOACH in the episode of care (% difference in Charges between JointCOACH and standard of care groups)

#### 4. Methods

#### 4.1 Study Design

The study design is a prospective, randomized trial in which patients undergoing elective primary hip or knee arthroplasty will be offered perioperative use of JointCOACH vs standard of care. A total of 400 patients will be enrolled (200 in each group). The following outcome measures will be collected at the intervals specified in the Schedule of Events:

- Demographics (Age, gender, BMI)
- Comorbidities (Age-Adjusted Charlson Comorbidity Index)
- Surgical details (ASA (or other comorbidity index), Length of surgery (incision to closure), procedure type, operative limb, surgeon)
- Length of hospital stay and discharge disposition
- Number of ED visits and follow-up visits within 90 days
- Number of phone calls and on-call pages within 90 days
- Readmissions and reoperations within 90 days
- Patient satisfaction (VAS satisfaction and PPE-15)
- Provider satisfaction (5-point Likert scale)

#### **4.2 Patient Population**

The Cleveland Clinic Orthopedic Institute practice patients from Main Campus surgeons (Mesko, Krebs, Greene, Kamath, Piuzzi), Lutheran Hospital surgeons (Mesko, Krebs), Marymount surgeons (Kamath, Piuzzi), and Medina Hospital surgeons (Greene) will be assessed for eligibility.

#### Inclusion criteria

- 1. Undergoing primary total hip or primary total knee arthroplasty
- 2. Willing to sign an IRB approved informed consent form
- 3. Have internet access or mobile access with a valid email address at the time of enrollment
- 4. Above the age of 18 years

#### Exclusion criteria

1. Staged arthroplasty procedure within 6 months of the index procedure

- 2. Abandoned email address of record (e.g. bounce of email from clinic)
- 3. Planned discharge to a Skilled Nursing Facility

#### **4.3 Sample Size Calculation**

We will enroll 400 patients (200 in each group). This sample size was estimated using patient reported satisfaction based on the PPE-15 questionnaire as the primary endpoint. Currently, it is not known what will be a clinically relevant difference so we conservatively estimated that a 10% difference in patient satisfaction (difference in % of respondents indicating a problem on the PPE-15 between treatment and control groups) would be relevant. Based on data published in a study by Jenkinson et al, we used a mean of 24.7% (± 7.7) for the percent of respondents across all PPE-15 domains that identified a problem with their experience<sup>6</sup>. Setting alpha equal to 0.05 and power equal to 80%, we determined that we will need 153 patients in each group. However, we will enroll 200 patients in each group to account for withdrawals and non-responders.

## 4.4 Schedule of Events

| <b>Evaluation</b> | Preop | Intraop | Inpatient | <u>D1</u> | <u>D2</u> | <u>D3</u> | <u>D4</u> | <u>D6</u> | <u>D8</u> | <b>D10</b> | D12 | W1-2 | W4-6 | <b>D30</b> | <b>D90</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Demographics | X | | | | | | | | | | | | | | |
| Medical History / Comorbidities | X | | | | | | | | | | | | | | |
| Surgical Details | | X | | | | | | | | | | | | | |
| Discharge (LOS, disposition) | | | X | | | | | | | | | | | | 1 |
| Track Readmission / Reoperation | | | | | | | | | | | | | | X | X |
| Track ED visits, office visits | | | | | | | | | | | | | | X | X |
| Track calls and on-call pages | | | | | | | | | | | | | | X | X |
| Adverse Events | | X | X | | | | | | | | | | | X | X |
| Postop Check-in Check-up | | | | X | X | X | X | X | X | X | X | | | | |
| Recovery Goals | | | | | | | | | | | | X | X | | |
| HOOS Jr / KOOS Jr | X | | | | | | | | | | | | | | X |
| Promise 10 | X | | | | | | | | | | | | | | X |
| Patient Satisfaction (VAS and PPE-15) | | | | | | | | | | | | | | X | X |
| Provider Satisfaction (5-point Likert) | | | | | | | | | | | | | | | X |

#### 4.5 Data Analysis Plan

The difference in percent of respondents indicating a problem on the PPE-15 between treatment and control groups will be calculated as [percent of standard of care respondents reporting a problem, averaged across all PPE-15 domains] – [percent of JointCOACH respondents reporting a problem, averaged across all PPE-15 domains], such that a positive difference indicates that the JointCOACH group was more satisfied than the standard of care group, while a negative value indicates the opposite. A superiority hypothesis test using the two-independent sample t-test will be used to statistically evaluate the difference in the average satisfaction between groups.

#### 5. References

- 1. Coulter A, Ellins J. Effectiveness of strategies for informing, educating, and involving patients. *BMJ*. 2007;335(7609):24-27. doi:10.1136/bmj.39246.581169.80.
- 2. Hibbard JH, Greene J, Overton V. Patients with lower activation associated with higher costs; delivery systems should know their patients' "scores". *Health Aff (Millwood)*. 2013;32(2):216-222. doi:10.1377/hlthaff.2012.1064.
- 3. Graarup J, Ferrari P, Howard LS. Patient engagement and self-management in pulmonary arterial hypertension. *Eur Respir Rev.* 2016;25(142):399-407. doi:10.1183/16000617.0078-2016.
- 4. Lee CS, Bidwell JT, Paturzo M, et al. Patterns of self-care and clinical events in a cohort of adults with heart failure: 1 year follow-up. *Heart Lung*. 2018;47(1):40-46. doi:10.1016/j.hrtlng.2017.09.004.
- 5. Ryu B, Kim N, Heo E, et al. Impact of an Electronic Health Record-Integrated Personal Health Record on Patient Participation in Health Care: Development and Randomized Controlled Trial of MyHealthKeeper. *J Med Internet Res.* 2017;19(12):e401. doi:10.2196/jmir.8867.
- 6. Jenkinson C, Coulter A, Bruster S. The Picker Patient Experience Questionnaire: development and validation using data from in-patient surveys in five countries. *Int J Qual Heal care J Int Soc Qual Heal Care*. 2002;14(5):353-358.

# 6. Appendix

# **6.1 Study Metrics**

| Metric | Justification |
|---|---|
| Patient Reported satisfaction – VAS and PPE-15 | -Substantial opportunity for the Cleveland Clinic to |
| | differentiate itself among health systems and enhance |
| | revenue associated with patient satisfaction measures |
| Patient utilization and compliance | - Substantial opportunity for national exposure as related |
| | to national directives to drive patient engagement (See |
| | NCQA's Leadership Series: Focus on Patient |
| | Engagement at |
| | http://www.qualityprofiles.org/leadership_series/patient |
| | _engagement/index_patient_engagement.asp) |
| Physician and staff satisfaction | - Opportunity to demonstrate clinical adoption rates and |
| | low barriers to implementation. |
| Total 90 day post-operative cost from index date+1 | Joint Coach templates should be able to either <i>prevent</i> |
| (same day) or from index date + LOS (inpatient)* | the complication, or through early detection at the clinic |
| *Claima = 1i4 = 1i4 :: 00 1 1 :: i4 = 1i4 | level, reduce expense through minimized emergency room visits and readmissions. |
| *Claims submitted within 90 days must be limited to | room visits and readmissions. |
| ICD-10 listed below (or if hospitalization due to ICD-10 below) in order to exclude unrelated claims. | |
| 30 day post-op hospitalization rate (this is a | |
| readmission if initially an inpatient procedure, or an | |
| admission if initially an outpatient procedure)* | |
| *Must be associated with ICD-10s listed below in | |
| order to exclude unrelated readmissions. | |
| 30-day ED Visit Rate* | |
| *Must be associated with ICD-10s listed below in | |
| order to exclude unrelated ED visits. | |
| Number of follow up visits within 90 days | Demonstration to physicians and practices the potential |
| The second of the second of th | to improve throughput and workflow efficiency by |
| | minimizing the number of follow up visits required. |
| Potentially preventable readmissions and | Potentially preventable admissions, events, ED visits. |
| complications identified using JointCOACH | Using an approach similar to 3M's Potentially |
| | Preventable Events grouping software, we will examine |
| | all events (ED visits, admissions, complications) for |
| | relation to index event, and compare this rate to prior |
| | year. Data may be supplemented by Physician survey. |
| | http://solutions.3m.com/wps/portal/3M/en_US/Health- |
| | Information-Systems/HIS/Products-and- |
| | Services/Products-List-A-Z/PPR-and-PPC-Grouping- |
| | Software/ |

## 6.2 ICD-10 codes for relevant metrics

| Description | ICD-10 |
|---|---|
| 1. Must be in 1st or 2nd diagnosis and must not be chronic, or | |
| 2. If patient is admitted, must be in 1st or 2nd diagnosis on hospital discharge. | |
| Infection and inflammatory reaction due to internal prosthetic device, implant, and graft | |
| <ul> <li>Due to unspecified implant, device, and graft</li> </ul> | |
| <ul> <li>Due to internal joint prosthesis</li> </ul> | T8579XA |
| <ul> <li>Due to other internal orthopedic device, implant and graft</li> </ul> | T8450XA |
| | T8460XA |
| Other complications of internal prosthetic device, implant, and graft | |
| <ul> <li>Due to unspecified implant, device, and graft</li> </ul> | T859XXA |
| • Due to internal joint prosthesis | T8481XA- |
| <ul> <li>Due to other internal orthopedic device, implant, and graft</li> </ul> | T8486XA; |
| | T8489XA;<br>T849XXA |
| | 1049AAA |
| Postoperative infection | |
| Other post-operative infection (abscess, septicemia) | K6811 |
| | T814XXA |
| Disruption of wound | |
| <ul> <li>Dehiscence of operation wound</li> </ul> | T8130XA- |
| | T8132XA |
| Infections of Skin and Subcutaneous Tissue | T. C. C. C. C. |
| Upper arm and forearm | LO3119 |
| <ul> <li>Leg except foot</li> </ul> | LO3129 |
| <ul> <li>Abscess NOS, Cellulitis NOS</li> </ul> | LO390 |
| | LO391 |
| Gastrointestinal hemorrhage | |
| Hematemesis | K920 |
| <ul> <li>Melena</li> </ul> | K921 |
| <ul> <li>Hemorrhage of gastrointestinal tract, unspecified</li> </ul> | K922 |
| Hemorrhage NOS | R58 |
| Venous embolism and thrombosis of deep vessels of lower extremity | I82409 |
| Of unspecified site | I8291 |
| Pulmonary embolism and infarction | I2690 |
| | 12692 |
| | 12699 |
| | T82817A, |
| | T82818A |
| Since ED coding is often not as precise as the above, we will likely need to also have | |
| these below | |
| Fever unspecified | R502 |
| | R509 |
| | R5081- |
| | R5094 |
| Creatomic inflammatows reamoned are drawn don't infectious accountillated to | R6883 |
| Systemic inflammatory response syndrome due to infectious process without acute organ dysfunction | A419 |
| Severe sepsis | R6520 |
| Joint Replacement DRGs | 461-462, |
| John Replacement DROS | 469-470 |
| Hip and Knee specific DRGs | 466-468, |
| Inp and Inico specific Bross | 488-489 |

# **6.3 Success Thresholds for Study Metrics**

| Metric | Threshold | Rationale |
|---|---|---|
| Patient reported () satisfaction | ≥ 70% satisfied or very satisfied | Value is consistent with most of the Medicare value based purchasing programs. 70% also exceeds thresholds targeted by several other large health systems. |
| Patient engagement | ≥ 70% of members are ≥ 60% engaged with the Joint Coach software | |
| Physician satisfaction | > 80% physician satisfaction | |
| Total 90 day post-operative cost (claims submitted) from index date+1 (same day) or from index date + LOS (inpatient) | No increase in cost during pilot study relative to cost averaged across 3 prior years (costs to be adjusted for inflation using either the medical care component of the Bureau of Labor Statistics Consumer Price Index, or The health system internal inflation index if available.) | Standard inflationary cost adjustment in medical economics is the medical care component of the CPI, or using a 3% discount rate. |
| 30-day post-op hospitalization rate | < 4% considering the UHC national average | |
| 30-day ED visit rate | | |
| Number of follow up visits within 90 days | | |
| Potentially preventable admissions | | |

# **Provider Satisfaction Survey**

| What is your role? | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| □ Surgeon | □ Phys | ician Assist | ant | □ Nurse | | | | | |
| How satisfied are you with the use of JointCOACH? | | | | | | | | | |
| □ Very Dissa | atisfied | ☐ Dissatis | sfied | □ Ne | utral | □ Sa | tisfied | □ Very S | Satisfied |
| How likely are you to recommend JointCOACH to others? | | | | | | | | | |
| □ Very Unlik | kely □ | l Unlikely | □N | eutral | □ Li | kely | □ Ver | y Likely | |